CLINICAL TRIAL: NCT03826433
Title: Clinical Study of Human Umbilical Cord Mesenchymal Stem Cells (19#iSCLife®-LC) in the Treatment of Decompensated Hepatitis b Cirrhosis
Brief Title: hUC Mesenchymal Stem Cells (19#iSCLife®-LC) in the Treatment of Decompensated Hepatitis b Cirrhosishepatitis b Cirrhosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sclnow Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCLnow-XY-04
Record Dates: First submitted 2019-01-14; First posted 2019-02-01 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Hepatitis B
Keywords: Hepatitis B Cirrhosis, mesenchymal stem cell
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Mesenchymal Stem Cells : through peripheral intravenous slowly, every time 6*10^7 (30ml) Other medication of Treatment Group: before the30min of first time to inject stem cells, Intravenous methylprednisone 20mg. All patients require oral nucleoside drugs resistant hepatitis B virus treatment.Use stem cell therapy, by Peripheral iv, 6 * 10 ^ 7 (30 ml)
  Interventions: Biological: Peripheral iv
- Control Group (No Intervention): Control Group: Using basic contrast .

INTERVENTIONS:
Biological: Peripheral iv — 6*10^7 cells
  Arms: Treatment Group

SUMMARY:
1. Evaluation the safety of using human umbilical mesenchymal stem cells to treat patients with hepatitis B cirrhosis.
2. Observe the curative effect of patients with hepatitis B cirrhosis who use human umbilical mesenchymal stem cells to treat.
3. Explore the possible mechanism of human umbilical mesenchymal stem cells to treat patients with hepatitis B cirrhosis.

DETAILED DESCRIPTION:
This experimental use umbilical cord mesenchymal stem cells in treatment of decompensated hepatitis B cirrhosis to evaluate its safety and efficacy,

This experimental is mainly aimed at people aged 18-60 years old, regardless of gender and with body mass index (BMI) between 19-25kg/m2 (including boundary value). It was decided into treatment group and control group to evaluate the effectiveness and safety of mesenchymal stem cells by peripheral intravenous injection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years old, gender not limited, body mass index (BMI) between 19-25 kg/m2, including boundary value;
* The diagnosis of hepatitis B cirrhosis was in line with the 2015 American society of hepatology (AASLD) guidelines for the treatment of chronic hepatitis B, and the liver function grade was child-pugh B or child-pugh C, with a score range of 7-12 points, and Model for End-Stage Liver Disease score≤21 points.
* Have not received stem cell therapy in the recent 6 months;
* Subjects will be able to sign the informed consent in accordance with the study procedures and instructions.

Exclusion Criteria:

* Insufficiency of vital organs, such as heart, kidney and lung;
* End-stage cirrhosis with severe complications, including but not limited to: hepatic encephalopathy, gastrointestinal bleeding,Severe bleeding tendency, massive ascites, etc.
* Concomitant peritonitis, pneumonia, or other types of infection not under control;
* Have a history of severe allergic reaction or allergy to two or more kinds of food or medicine;
* Positive serum HIV antibody and syphilis antibody;
* Alpha fetoprotein>400ng/mL with primary liver cancer or without imaging evidence;
* Chronic liver disease and cirrhosis are caused by non-chronic hepatitis B virus infection, or other factors except chronic hepatitis B virus infection ;
* Patients with severe mental illness and cognitive impairment;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Validity evaluation by detection of the Model for end-stage Liver Disease score of participants | 12 month
  After finish the mesenchymal stem cell treatment, observe the change in baseline outcome measures.
  40 or more - 71.3% observed mortality 30-39 - 52.6% observed mortality 20-29 - 19.6% observed mortality 10-19 - 6.0% observed mortality <9 - 1.9% observed mortality

SECONDARY OUTCOMES:
Safety evaluation by detecting Blood routine | 12 month
  To calculate the number of hemocyte and related protein (e.g. erythrocyte, lymphocyte, and hemoglobin) after mesenchymal stem cell treatment
Validity evaluation by detection of the child-pugh of participants | 12 month
  After finish the mesenchymal stem cell treatment, observe the change in baseline outcome measures.
  Points Class One-year survival Two-year survival 5-6 A 100% 85% 7-9 B 80% 60% 10-15 C 45% 35%

OTHER OUTCOMES:
Validity evaluation by detection of the coagulation function of participants | 12 month
  After finish the mesenchymal stem cell treatment, observe the change of Prothrombin Time and International Normalized Ratio (PT/INR) in baseline outcome measures.
  The time is around 12-13 seconds, the INR in absence of anticoagulation therapy is 0.8-1.2.
Imaging examination | 12 month
  After finish the mesenchymal stem cell treatment, observe the Computed Tomography (CT).
Imaging examination | 12 month
  Fibro-Touch examination
Safety evaluation by detecting adverse events and serious adverse events | 12 month
  To evaluate the changes of safety indexes before and after mesenchymal stem cell treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xuegong Fan, doctor, Study Director — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No